CLINICAL TRIAL: NCT01142180
Title: Early Selective Angiographic Embolization to Severely Bleeding Peptic Ulcers After Their Initial Endoscopic Hemostasis - a Randomized Controlled Trial
Brief Title: Early Selective TAE to Severely Bleeding Peptic Ulcers After Their Initial Endoscopic Hemostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAE2
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Bleeding; Peptic Ulcer; Arterial Embolization
Keywords: Bleeding peptic ulcer; Active bleeding; Trans-arterial angiographic embolization
MeSH Terms: conditions — Hemorrhage; Peptic Ulcer; Peptic Ulcer Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAE group (Active Comparator): Patients will be undergone TAE after endoscopic hemostasis.
  Interventions: Procedure: TAE
- No TAE group (Active Comparator): No TAE procedure will be performed after endoscopic treatment.
  Interventions: Procedure: No TAE

INTERVENTIONS:
Procedure: TAE — The procedure will be performed within 12 hours of endoscopic therapy. This is usually performed under conscious sedation
  Other Names: Transarterial embolization
  Arms: TAE group
Procedure: No TAE — No TAE procedure will be performed after endoscopic treatment
  Arms: No TAE group

SUMMARY:
The aim of this study is to determine if early angiographic embolization can forestall recurrent bleeding in selected high risk ulcers after their initial endoscopic control; to validate prospectively the investigators proposed in selecting high risk ulcers for recurrent bleeding in spite of maximal endoscopic control and profound acid suppression using high dose intravenous infusion of proton pump inhibitor; to characterize the nature of bleeding arteries in severely bleeding peptic ulcers and determine the efficacy of angiographic embolization in the prevention of recurrent bleeding and to establish safety profile of angiographic embolization as an early elective treatment to bleeding peptic ulcers.

DETAILED DESCRIPTION:
Endoscopic therapy is now the treatment of choice in patients with actively bleeding peptic ulcers and ulcers with non-bleeding visible vessels. Following endoscopic control of bleeding, we showed that the use of a high dose intravenous infusion of proton pump inhibitor (PPI) for 72 hours further reduced rate of recurrent bleeding [Lau NEJM 2000]. Recurrent bleeding still occurs in 8 to 10 percent of patients who receive the above treatment regime. The associated mortality following a rebleed is 4-10 fold higher when compared to those without recurrent bleeding. In a logistic regression model involving 1144 patients after successful endoscopic thermocoagulation to their bleeding peptic ulcers, we demonstrated that several factors independently predicted recurrent bleeding. They included hypotension, hemoglobin <10g/dl, fresh blood in the stomach, ulcer size > 2cm and active bleeding during endoscopy [Wong Gut 2003]. When we applied this model in a cohort of 945 patients who underwent endoscopic control of bleeding to their ulcers and adjunctive use of high dose intravenous PPI, 275 belonged to the high risk group. Of them, rebleeding leading to surgery or death occurred in 46 patients (16.7%)[Chiu DDW 2007]. Endoscopic treatment to bleeding peptic ulcers has its own limit. In an ex vivo bleeding model using canine mesenteric arteries, endoscopic thermocoagulation could only consistently seal arteries up to 2 mm in size [Johnson Gastro 1987]. Trans-arterial angiography allows clinicians to study and characterize bleeding arteries underneath peptic ulcers. In ulcers that erode into major arteries such as the gastro-duodenal artery complex and branches from left gastric artery, angiography complements endoscopic therapy in the form of selective coiling of the bleeding artery. Trans-arterial angiographic coiling can provide definitive control of bleeding from larger arteries i.e. > 2 mm in size. In cohort studies, trans-arterial angiographic coiling has been shown to compare favorably to surgery, and is less invasive in the control of severe bleeding in peptic

ELIGIBILITY:
Inclusion Criteria:

* Actively bleeding peptic ulcers (Forrest I), NBVV or Forrest IIa ulcer,
* Successful endoscopic hemostasis by combination treatment of injected epinephrine followed by either 3.2mm heat probe 30J (4 continuous pulses) or hemo-clipping (at least 2 clips) And one of the followings
* Spurting hemorrhage during endoscopy;
* Ulcer >= 2 cm is determined by an opened biopsy forceps;
* Hb on admission of < 9 g/dl; or
* Hypotension prior to endoscopy defined by SBP of <90 mmHg AND HR of >110 bmp

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
clinical re-bleeding | within 30 days of therapy
  Clinical rebleeding is defined by fresh hematemesis, fresh melena or hematochezia and signs of hypovolemic shock (systolic blood pressure of <90mmHg and pulse rate >110 per minute) and a drop in hemoglobin of > 2 g/dl per 24 hours despite adequate transfusion.
  Rebleeding will be confirmed by an immediate endoscopy showing fresh blood in stomach or active bleeding from a previously seen ulcer. A clinical rebleeding will be independently reviewed by an adjudication panel.

SECONDARY OUTCOMES:
death from all causes | within 30 days of therapy
  death from all causes
transfusion requirement | within 30 days of therapy
  transfusion requirement
hospital stay including Intensive Care Unit stay | within 30 days of therapy
  hospital stay including Intensive Care Unit stay
further interventions either further TAE or surgery | within 30 days of therapy
  further interventions either further TAE or surgery
hospital costs | within 30 days of therapy
  hospital costs

CONTACTS AND LOCATIONS:
Overall Officials: James Y LAU, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Derived] Lau JYW, Pittayanon R, Wong KT, Pinjaroen N, Chiu PWY, Rerknimitr R, Holster IL, Kuipers EJ, Wu KC, Au KWL, Chan FKL, Sung JJY. Prophylactic angiographic embolisation after endoscopic control of bleeding to high-risk peptic ulcers: a randomised controlled trial. Gut. 2019 May;68(5):796-803. doi: 10.1136/gutjnl-2018-316074. Epub 2018 May 25. PMID 29802172